CLINICAL TRIAL: NCT01663298
Title: FGF2 Promoter Hypermethylation and Implant Wound Healing Among Smokers and Diabetics
Brief Title: Gene Expression Variation and Implant Wound Healing Among Smokers and Diabetics
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10-1184; 1R01DE021052-01 (NIH); 1UL1RR025747 (NIH); AWU (Other: UNC)
Record Dates: First submitted 2012-08-01; First posted 2012-08-13 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2019-02

CONDITIONS: Smoking; Diabetes
Keywords: DNA methylation; FGF2; Wound healing; Smoking; Diabetes; Implant
MeSH Terms: conditions — Smoking; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Gingival tissues, gingival crevicular fluid, saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control group: Subjects must have never smoked and must be non-diabetic.
  Interventions: Procedure: Dental implant surgery
- Smoking group: Subjects must have had at least 5 pack-years of self-reported smoking history, must be currently smoking and must be non-diabetic.
  Interventions: Procedure: Dental implant surgery
- Diabetic group: Subjects must have type 2 diabetes. The condition must be diagnosed subjects must be treated by medications and/or insulin. A HbA1C test result either within past 3 months or performed in the first visit must be available. They must have never smoked.
  Interventions: Procedure: Dental implant surgery

INTERVENTIONS:
Procedure: Dental implant surgery — Surgery involving placement of one dental implant, of either Astra Tech or Straumann system, is performed in all subjects within 2 weeks of screening examination. Implant placement is 1-stage, but can be either on edentulous ridges or in extraction sockets.This is not a randomized treatment arm/group design. The study is observational with regards to the analysis of tissue samples that are collected prior to the routine placement of implants. The implant choice is based upon patient needs and is not related to any outcome.

SUMMARY:
Periodontal wound healing is a complex multifactorial process that involves interactions among various cells, growth factors, hormones and extracellular matrices. Although still poorly understood, these interactions trigger a series of events that lead to new tissue formation. One growth factor that plays an important role in wound healing is fibroblast growth factor 2 (FGF2). Many animal and human studies have shown this protein is effective in periodontal regeneration. Recently, epigenetic modifications, such as DNA methylation, have been associated with changes in patterns of gene expression. Preliminary data suggests that FGF2 gene may be differentially methylated in periodontal tissues. Aberrant gene promoter methylation in smokers and diabetics has also been reported in many studies. However, the role of DNA methylation in wound healing has not yet been investigated.

The investigators hypothesize that the methylation status of FGF2 gene can affect the levels of FGF2 secreted during wound healing phase after dental implant surgery. The investigators also hypothesize there exists a difference in methylation levels of FGF2 gene in healthy, smoking and diabetic patients that can interfere with wound healing. The investigators seek to determine whether DNA methylation plays a role in wound healing and whether the methylation level of FGF2 gene varies among healthy, smoking and diabetic patients.

DETAILED DESCRIPTION:
Periodontal wound healing is a complex multifactorial process that involves interactions among various cells, growth factors, hormones and extracellular matrices. Although still poorly understood, these interactions trigger a series of events that lead to new tissue formation. One growth factor that plays an important role in wound healing is fibroblast growth factor 2 (FGF2). FGF2 is a member of the heparin-binding growth factor family, secreted by macrophages and endothelial cells. During the proliferative healing phase, it stimulates fibroblast proliferation & ECM synthesis, and increases chemotaxis, proliferation and differentiation of endothelial cells. During the bone remodeling phase, FGF2 also stimulates mesenchymal progenitor cell migration. Many animal and human studies have shown FGF2 are effective in periodontal regeneration. In 1999, Murakami showed surgically treated 3-wall intrabony defect in dogs grafted with FGF2 was able to demonstrate significantly greater cementum and bone formation. Four years later, his group again found that topical application of rhbFGF in surgically treated class 2 furcation defects in dogs also showed increase in formation of PDL, cementum and bone. In 2008, Kitamura performed a randomized controlled study in humans with 2- or 3-wall intrabony periodontal defects and found that rhbFGF was able to stimulate alveolar bone growth and PDL regeneration.

Recently, epigenetic modifications, such as DNA methylation, have been associated with changes in patterns of gene expression that do not involve changes in DNA sequence. DNA methylation is characterized by the addition of the methyl group onto cytokines within CpG regions. Methylated CpG regions interfere with the access of transcription factors to the promoter region, thereby silencing the gene. This DNA methylation phenomenon has important regulatory functions in normal and pathological cellular processes. It was recognized that alteration in the methylation states at the promoter regions of tumor suppressor genes are implicated with cancer. A persistent inflammation was also observed to cause DNA methylation, which inactivates suppressors of cytokine signaling and results in exaggerated cytokine production. This makes an individual susceptible to periodontal disease. In our laboratory, the investigators have discovered that periodontal disease is associated with increased DNA methylation of the COX-2 promotor, especially the locus immediately adjacent to the NF-kB in the promoter region. Preliminary data (not shown) suggests that FGF2 may be differentially methylated in periodontal tissues. Aberrant gene promoter methylation in smokers and diabetics has also been reported in many studies. However, the role of DNA methylation in wound healing has not yet been investigated.

We hypothesize that the methylation status of FGF2 can affect the levels of FGF2 secreted during wound healing phase after dental implant surgery. We also hypothesize there exists a difference in methylation levels of FGF2 in healthy, smoking and diabetic patients that can interfere with wound healing. We seek to determine whether DNA methylation plays a role in wound healing and whether the methylation level of FGF2 varies among healthy, smoking and diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females between the age of 18 and 70 years (inclusive)
* Able and willing to follow study procedures and instructions
* Have read, understood and signed an informed consent form
* In good general health
* Have one or more implant placements as their future treatment needs. The implant placement can be either as one-stage or two-stage, and can be either in an edentulous ridge or an extraction socket
* Qualify for enrollment into one of the three study groups
* Have probing depth ≤ 4 mm for all teeth at the same quadrant of implant placement. Sites with probing depth 5 mm will also be included if bleeding on probing in these sites are absent.

Exclusion Criteria:

* Have a chronic disease with oral manifestations
* Exhibit gross oral pathology
* Use of either antibiotics or NSAIDs within 1 month prior to screening examination
* Chronic treatment (i.e. two weeks or more) with any medication known to affect periodontal status (e.g. phenytoin, calcium, antagonists, cyclosporin, Coumadin) within 1 month prior to screening examination
* Systemic conditions, except smoking and diabetes, that are known to affect the periodontal status
* With active infectious diseases such as hepatitis, HIV or tuberculosis
* Known to be pregnant or breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients in the graduate periodontal clinic in the school of dentistry at the University of North Carolina
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2010-08; Primary Completion 2016-01-12 (Actual); Study Completion 2016-02-23 (Actual)

PRIMARY OUTCOMES:
FGF2 methylation level | On the day of implant surgery
  Genomic DNA is isolated from the collected gingival tissue samples. Methylation alterations in FGF2 are detected through differential methylation hybridization using the EpiTect® Methyl qPCR single assay.

SECONDARY OUTCOMES:
FGF2 mRNA expression level | On the day of implant surgery (DAY 0)
  RNA is isolated from the collected gingival tissue samples and is then processed for gene expression analysis by quantitative real-time PCR.
FGF2 protein level | On the day of implant surgery (DAY 0) and 2, 4 and 6 weeks following implant surgery
  Gingival crevicular fluid, obtained from the two adjacent sites closest to the implant location, is used to quantify specific FGF2 protein levels by ELISA.
Implant stability quotient (ISQ) | 4 and 6 weeks following implant surgery
  The degree of implant stability at various time points following the surgery is measured using an Osstell ISQ instrument. An ISQ value, ranged between 1 and 100, is generated for each sample at each time point.
Wound healing indices (WHI) | 2, 4 and 6 weeks following implant surgery
  The degree of soft tissue healing at various time points following surgery is monitored by WHI.

CONTACTS AND LOCATIONS:
Overall Officials: Silvana Barros, DDS, PhD, MS, Principal Investigator — UNC Chapel Hill School of Dentistry
Locations (1):
- Department of Periodontology, UNC School of Dentistry, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Kaigler D, Cirelli JA, Giannobile WV. Growth factor delivery for oral and periodontal tissue engineering. Expert Opin Drug Deliv. 2006 Sep;3(5):647-62. doi: 10.1517/17425247.3.5.647. PMID 16948560
- [Background] Murakami S, Takayama S, Ikezawa K, Shimabukuro Y, Kitamura M, Nozaki T, Terashima A, Asano T, Okada H. Regeneration of periodontal tissues by basic fibroblast growth factor. J Periodontal Res. 1999 Oct;34(7):425-30. doi: 10.1111/j.1600-0765.1999.tb02277.x. PMID 10685372
- [Background] Murakami S, Takayama S, Kitamura M, Shimabukuro Y, Yanagi K, Ikezawa K, Saho T, Nozaki T, Okada H. Recombinant human basic fibroblast growth factor (bFGF) stimulates periodontal regeneration in class II furcation defects created in beagle dogs. J Periodontal Res. 2003 Feb;38(1):97-103. doi: 10.1034/j.1600-0765.2003.00640.x. PMID 12558943
- [Background] Kitamura M, Nakashima K, Kowashi Y, Fujii T, Shimauchi H, Sasano T, Furuuchi T, Fukuda M, Noguchi T, Shibutani T, Iwayama Y, Takashiba S, Kurihara H, Ninomiya M, Kido J, Nagata T, Hamachi T, Maeda K, Hara Y, Izumi Y, Hirofuji T, Imai E, Omae M, Watanuki M, Murakami S. Periodontal tissue regeneration using fibroblast growth factor-2: randomized controlled phase II clinical trial. PLoS One. 2008 Jul 2;3(7):e2611. doi: 10.1371/journal.pone.0002611. PMID 18596969
- [Background] Barros SP, Offenbacher S. Epigenetics: connecting environment and genotype to phenotype and disease. J Dent Res. 2009 May;88(5):400-8. doi: 10.1177/0022034509335868. PMID 19493882
- [Background] Gomez RS, Dutra WO, Moreira PR. Epigenetics and periodontal disease: future perspectives. Inflamm Res. 2009 Oct;58(10):625-9. doi: 10.1007/s00011-009-0041-7. Epub 2009 May 8. PMID 19440658
- [Background] Wilson AG. Epigenetic regulation of gene expression in the inflammatory response and relevance to common diseases. J Periodontol. 2008 Aug;79(8 Suppl):1514-9. doi: 10.1902/jop.2008.080172. PMID 18673005
- [Background] Ling C, Groop L. Epigenetics: a molecular link between environmental factors and type 2 diabetes. Diabetes. 2009 Dec;58(12):2718-25. doi: 10.2337/db09-1003. No abstract available. PMID 19940235
- [Background] Krupanidhi S, Sedimbi SK, Vaishnav G, Madhukar SS, Sanjeevi CB. Diabetes--role of epigenetics, genetics, and physiological factors. Zhong Nan Da Xue Xue Bao Yi Xue Ban. 2009 Sep;34(9):837-45. PMID 19779253
- [Background] Simmons RA. Developmental origins of diabetes: the role of epigenetic mechanisms. Curr Opin Endocrinol Diabetes Obes. 2007 Feb;14(1):13-6. doi: 10.1097/MED.0b013e328013da5b. PMID 17940413
- [Background] Kuroda A, Rauch TA, Todorov I, Ku HT, Al-Abdullah IH, Kandeel F, Mullen Y, Pfeifer GP, Ferreri K. Insulin gene expression is regulated by DNA methylation. PLoS One. 2009 Sep 9;4(9):e6953. doi: 10.1371/journal.pone.0006953. PMID 19742322
- [Background] Han W, Wang T, Reilly AA, Keller SM, Spivack SD. Gene promoter methylation assayed in exhaled breath, with differences in smokers and lung cancer patients. Respir Res. 2009 Sep 25;10(1):86. doi: 10.1186/1465-9921-10-86. PMID 19781081
- [Background] Belinsky SA, Palmisano WA, Gilliland FD, Crooks LA, Divine KK, Winters SA, Grimes MJ, Harms HJ, Tellez CS, Smith TM, Moots PP, Lechner JF, Stidley CA, Crowell RE. Aberrant promoter methylation in bronchial epithelium and sputum from current and former smokers. Cancer Res. 2002 Apr 15;62(8):2370-7. PMID 11956099